CLINICAL TRIAL: NCT00812292
Title: A Phase I, Open-label, Randomized, Crossover Trial in Healthy Adults to Compare the Oral Bioavailability of TMC278 From Three Concept Pediatric Formulations (Solution, Suspension, Granules) With That From the Adult Phase III Tablet Formulation.
Brief Title: TMC278-TiDP38-C145: A Bioavailability Study in Healthy Adult Volunteers to Evaluate 3 Pediatric Formulations of TMC278 (a Solution, a Suspension, and Granules) Compared to an Adult Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR012586
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-04

CONDITIONS: Pharmacokinetics; Bioavailability; HIV-1
Keywords: TMC278; TMC278-C145; TMC278-TiDP38-C145; concept pediatric formulations of TMC278; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Rilpivirine

INTERVENTIONS:
Drug: TMC278

SUMMARY:
The purpose of this study is to evaluate how much and how fast a single, oral, daily 25 mg dose of TMC278 is absorbed into the body when administered as a solution, suspension, granules, or a tablet. In addition, the effect of each formulation of TMC278 will be evaluated in patients in the fasted and fed states and the palatability (how the drug tastes) of each formulation will be assessed. Finally, the safety and tolerability of each formulation of TMC278 will be assessed throughout the study.

DETAILED DESCRIPTION:
This is an open-label (both investigator and volunteer knows the name of the assigned study medication), randomized (study medication will be assigned by chance) cross-over study in healthy adults to compare the rate and the extent of absorption of TMC278 when administered as a single 25 mg dose of the 3 concept pediatric formulations (solution [10 mg/mL], suspension [5 mg/mL], granules [2.5 mg/g]), under fed and fasted conditions, to that when administered as the 25 mg TMC278 Phase III tablet formulation, under fed conditions, in healthy adults and to assess the effect of food on the bioavailability of TMC278 after a single 25 mg dose of the concept pediatric TMC278 formulations in healthy adults. The palatability of the 3 concept formulations will be assessed in a fasted state by use of a questionnaire and a visual analog scale. The short-term safety and tolerability of TMC278 following administration of 3 single oral doses of 25 mg, formulated as one of the concept pediatric formulations (under fed and fasted conditions) and as the Phase III tablet (under fed conditions), in healthy adults will be evaluated. TMC278 25 mg formulated as a solution, suspension, granules, or tablet will be administered orally (by mouth). Each volunteer will receive on the first day of one treatment session one TMC278 25 mg tablet. On the first day of the other sessions they receive a single dose of TMC278 25 mg formulated as a the solution, a suspension or granules.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection
* A Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Informed Consent Form signed voluntarily before the first trial-related activity
* Able to comply with protocol requirements
* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, electrocardiogram, vital signs, and the results of blood biochemistry and hematology tests and a urinalysis carried out at screening.

Exclusion Criteria:

* A positive HIV-1 or -2 test at trial screening
* Female, except if postmenopausal since more than two years, or post-hysterectomy or post-tubal ligation (without reversal operation)
* One or more risk factors for QTc prolongation
* Currently active gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory or infectious disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
For each treatment session, full pharmacokinetic profiles will be measured up to 168 hours post-dosing

SECONDARY OUTCOMES:
Safety and tolerability will be monitored throughout the trial. Palatability of the 3 concept formulations will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: Phase I, open-label, randomized, crossover trial in healthy adults to compare the bioavailability of 3 concept pediatric formulations of TMC278 to the adult 25 mg Phase III tablet formulation, and to assess the food effect for each concept formulation. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1005&filename=CR012586_CSR.pdf